CLINICAL TRIAL: NCT01603485
Title: Open-Label, Randomized, Crossover Study to Estimate the Pharmacokinetics, Bioavailability and Effect of Food on Single Dose Modified-Release Lersivirine (UK-453,061) 500 mg in Healthy Subjects
Brief Title: Study to Estimate the Pharmacokinetics, Bioavailability and Effect of Food on Single Dose Modified-release Lersivirine 500 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5271050
Record Dates: First submitted 2012-05-10; First posted 2012-05-22 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Healthy Volunteer
Keywords: Bioavailability; Pharmacokinetics; Lersivirine; Modified-release

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lersivirine (Experimental)
  Interventions: Drug: Lersivirine Immediate-Release (fasted); Drug: Lersivirine Modified-Release #1 (fasted); Drug: Lersivirine Modified-Release #2 (fasted); Drug: Lersivirine Modified-Release #3 (fasted); Drug: Lersivirine Modified-Release (fed)

INTERVENTIONS:
Drug: Lersivirine Immediate-Release (fasted) — Single 500 mg dose of Lersivirine Immediate-Release Tablets (2 x 250 mg)
Drug: Lersivirine Modified-Release #1 (fasted) — Single 500 mg dose of Lersivirine Modified-Release Tablet #1
Drug: Lersivirine Modified-Release #2 (fasted) — Single 500 mg dose of Lersivirine Modified-Release Tablet #2
Drug: Lersivirine Modified-Release #3 (fasted) — Single 500 mg dose of Lersivirine Modified-Release Tablet #3
Drug: Lersivirine Modified-Release (fed) — Single 500 mg dose of Lersivirine Modified-Release Tablet dosed with food.

SUMMARY:
The purpose of this study is to estimate the pharmacokinetics (PK) of 3 different modified-release formulations of lersivirine and compare it to the PK of the immediate-release tablet. The effect of food on the PK of one of the modified-release tablets will also be assess along with the safety and tolerability of each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening;
* Treatment with an investigational drug within 60 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication;
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Lersivirine Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose
Lersivirine Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose
Lersivirine Maximum Observed Plasma Concentration (Cmax) | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose

SECONDARY OUTCOMES:
Lersivirine Plasma Decay Half-Life (t1/2) | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose
Lersivirine Time to Reach Maximum Observed Plasma Concentration (Tmax) | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose
Lersivirine Observed Plasma Concentration at time 24hr (C24) | T = 24 hours post dose
Lersivirine Last Observed Plasma Concentration (Clast) | T = 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 36 and 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271050&StudyName=Study%20to%20Estimate%20the%20Pharmacokinetics%2C%20Bioavailability%20and%20Effect%20of%20Food%20on%20Single%20Dose%20Modified-release%20Lersivirine%20500%20mg%20in%20Healthy